CLINICAL TRIAL: NCT03934593
Title: Building a Healthy Temple: a Diabetes Self-management Support Program in Hispanic Faith Community Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas at San Antonio (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Dr. Meizi He, Professor, The University of Texas at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ADA#1-17-ICTS-029
Record Dates: First submitted 2019-03-27; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Type2 Diabetes Mellitus
Keywords: diabetes; Hispanics; HbA1c; Self-Management Support Program
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: We will conduct a cluster randomized trial with repeated measures to compare the effectiveness of BHT DSMS intervention strategies among 360 adult diabetic congregants from 18 predominantly Hispanic churches in San Antonio, Texas (20 participants/church).
Who Masked: Participant
Masking Description: Using cluster randomized trial design; nine churches will be randomly assigned to the FB intervention (BHT DSMS), and nine to the FP intervention (Stanford DSMP).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faith-Based (FB, BHT DSMS) (Experimental): The BHT DSMD intervention strategies adapted Stanford DSMP in a spiritual context is used in this group. Participants in the FB group will participate in BHT DSMS, which includes a Health Sermon, a 6-session Health Bible Study with cooking demonstrations, the Stanford DSMP and a Diabetes Resource Seminar delivered by two trained church lay leaders.
  Interventions: Behavioral: Faith-Based (FB, BHT DSMS)
- Faith-Placed (FP, Stanford DSMP) (Active Comparator): The traditional Stanford DSMP is conducted in this control group. Participants in the FP group will first attend a 7-session community health and safety curriculum as a partial attention control intervention, followed by the Stanford DSMP and Diabetes Resource Seminar facilitated by the local public health department.
  Interventions: Other: Faith-Placed (FP, Stanford DSMP)

INTERVENTIONS:
Behavioral: Faith-Based (FB, BHT DSMS) — BHT DSMS Intervention components include Health Sermon and a 6-session Health Bible Study with cooking demonstrations, followed by the Stanford DSMP and a Diabetes Resource Seminar. All intervention activities are implemented by trained church lay leaders.
  Arms: Faith-Based (FB, BHT DSMS)
Other: Faith-Placed (FP, Stanford DSMP) — Standard Stanford DSMP delivered by health professional
  Arms: Faith-Placed (FP, Stanford DSMP)

SUMMARY:
The present study proposes to test the effectiveness of the Building a Healthy Temple: Diabetes Self-Management Support Program (BHT DSMS), a rendition of the Stanford DSMP in a spiritual context for the Hispanic faith community members. Using a holistic approach through integrating spiritual and physical health, BHT translates the Stanford DSMP in a way that may result in lasting behavior changes and improved diabetes outcomes for Hispanics with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The present study is proposing a 12-month translational study BHT DSMS to test the effectiveness of adapted Stanford DSMP in a spiritual context. A cluster randomized trial with repeated measures will be conducted to compare the effectiveness of DSMS intervention strategies among 360 adult diabetic congregants from 18 predominantly Hispanic churches in San Antonio, Texas (20 participants/church). Using cluster randomized trial design; nine churches will be randomly assigned to the Faith-Based (FB) intervention, and nine to the Faith-Placed (FP) intervention. The study will be implemented in two cohorts (8 churches for cohort 1 & 10 churches for cohort 2). All intervention activities will be implemented over 14 consecutive weeks. Participants in the FB group will participate in BHT DSMS, which includes a Health Sermon, a 6-session Health Bible Study with cooking demonstrations, the Stanford DSMP and a Diabetes Resource Seminar delivered by two trained church lay leaders. Participants in the FP group will first attend a 7-session community health and safety curriculum as a partial attention control intervention, followed by the Stanford DSMP and Diabetes Resource Seminar facilitated by the local public health department. The primary outcome will be a change in HbA1c levels. Secondary outcomes include: changes in body mass index (BMI), waist circumference (WC), quality of life, diabetes self-care behaviors, eating behavior and physical activity level. Data will be collected at baseline, 6, 9, and 12-months during the study period. The aims of present study are 1) To test feasibility of the Stanford DSMP in FP and FB settings through observation and documentation of the implementation process, in-depth interviews with program staff and focus groups with participants to identify facilitators and barriers of the intervention. 2) To translate Stanford DSMP in a spiritual context for Hispanic faith community members and compare the effectiveness of a FB versus FP approach in improving diabetes outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Church eligibility: [Churches must be predominantly Hispanics (60%) with at least 20 adult congregants with T2D willing to participate in the study. The rationale for 20 diabetic voluntary participants per church is based on the Stanford requirement of 12-16 participants allowed per support group and with an anticipated 25% attrition.]
* Participants' eligibility: Participants will be adults age 21 and above that have been diagnosed with T2D.

Exclusion Criteria:

* Children, adults under 21 years of age, and pregnant women

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
The change in HbA1c | Data is collected at baseline, 6, 9, and 12-months during the study period.
  A finger-prick blood sample will be collected for HbA1c testing using Metrika A1cNowTM (Bayer Health Care).

SECONDARY OUTCOMES:
Waist circumference | Data is collected at baseline, 6, 9, and 12-months during the study period.
  waist circumference (WC) will measured in the horizontal plane midway between the lowest rib and the iliac crest.
Body Mass Index | Data is collected at baseline, 6, 9, and 12-months during the study period.
  Participants' body weight and height will be measured. BMI will be calculated height and weight (kg/M2)
Quality of Life (QoL) | Data is collected at baseline, 6, 9, and 12-months during the study period.
  Quality of life in present study will be measured using the Problem Areas in Diabetes (PAID) scale (Polonsky and Anderson, 1995). The PAID measure of diabetes related emotional distress correlates with measures of related concepts such as depression, social support, health beliefs, and coping style, as well as predicts future blood glucose control of the patient. Questionnaire scale scoring: Each question has 5 possible answers with a value from 0 to 4, with 0 representing "no problem" and 4 "a serious problem". The scores are added up and multiplied by 1.25, generating a total score between 0 - 100. Patients scoring 40 or higher may be at the level of "emotional burnout" and warrant special attention. PAID scores in these patients may drop 10-15 points in response to
Diabetes Self-care practices | Data is collected at baseline, 6, 9, and 12-months during the study period.
  The Revised Summary of Diabetes Self-Care Activities (SDSCA) (Toobert, Hampson, and Glasgow, 2000). It is a 25-item self-report measure of the frequency of performing diabetes self-care tasks over the preceding 7 days. The response is based on a seven-point Likert scale to answer the question phrased as "On how many of the last 7 days did you…?". Higher overall scores reflect good diabetes self-care practice.
The barriers to diabetes care. | Data is collected at baseline, 6, 9, and 12-months during the study period.
  The barriers to diabetes care are investigated using selected questions from the National Survey of People with Diabetes (Harris, McGee, and Andrews, 2007).
Physical Activity (PA) level assessment | Data is collected at baseline, 6, 9, and 12-months during the study period.
  A 6-item Exercise Behaviors scale (Lorig et al 1996) measures total minutes per week of aerobic and nonaerobic exercise specifically over the past seven days. The first question measures the amount of time that the participant stretched or engaged in any strengthening exercises. The other five questions measures aerobic activity. The options for the questions include none, less than 30 minutes per week, 30-60 minutes per week, 1-3 hours per week, and more than 3 hours per week. The total aerobic and stretching and/or strengthening minutes were calculate by converting the "None" category to 0 minutes; "Less than 30 minutes/week" into 15 minutes; "30-60 minutes/week" into 45 minutes; "1-3 hours/week" into 120 minutes; and "More than 3 hours/week" into 180 minutes.(6) The response to the first question was used to determine the amount of time for stretching/strengthening while questions 2 through 6 were summed together to determine the amount of aerobic time.
Occupational physical activity | Data is collected at baseline, 6, 9, and 12-months during the study period.
  Occupational physical activity also is evaluated using a single-item question recommended by Behavioral Risk Factor Surveillance System (BRFSS) which is designed to categorize occupational physical activity into three components: 1) mostly sitting and standing (inactivity and low-intensity activity); 2) mostly waling (moderate-intensity activity); or 3) mostly heavy labor (vigorous-intensity activity) (www.cdc.gov/brfss/; Yore MM, Bowles HR, 2006)

OTHER OUTCOMES:
Diabetes self-efficacy | Data is collected at baseline, 6, 9, and 12-months during the study period.
  Diabetes self-efficacy scale will assess participants' diabetes self-efficacy (Sarkar, Fisher and Schillinger, 2006). It is an 8-item instrument assessing diabetic individual's self-management efficacy. These items addressed diabetes-specific domains such as confidence in self-monitoring of blood glucose (SMBG), as well as general health domains such as confidence in ability to get medical attention and take care of health using 4-point Likert-scale with responses from "1 = not at all sure" to "4 = very sure." For each item patients rated their confidence in their ability to perform a recommended self-care routine. The overall self-efficacy score are transformed to a 100-point scale with a higher score representing greater self-efficacy.
Social support in a spiritual context | Data is collected at baseline, 6, 9, and 12-months during the study period.
  Social support in a religion context will be measured using the instrument by Olphen et al.(2003) that assess the frequency with which participants receive support from other church members by asking "How often do people in your church or place of worship help you out? The answer options include "1= never; 2= hardly ever; 3= not too often; 4= fairly often and 5= very". Higher scores indicate greater levels of level of support.
Social support for diabetes self-management | Data is collected at baseline, 6, 9, and 12-months during the study period.
  • Social support for self-management will be assessed using modified Social Support Scale for Self-care in Middle-aged patients with type II diabetes (S4-MAD) (Naderimagham S, Niknami S, 2012) The questions in S4-MAD will be re-classified to evaluate the social support in emotional and information support, tangible support, affectionate support, positive support and additional support (www.rand.org). The social support resources include "Are you attending worship service at this church?", "Who help you the most in caring for your diabetes outside of church?", "Who helps you the most I caring for your diabetes within the church?". The responses will be "1 = Never; 2 = Rarely; 3 = Sometimes; 4 = Often; 5 = Always". The higher score reflects better spiritual coping.
Spiritual coping | Data is collected at baseline, 6, 9, and 12-months during the study period.
  Spiritual coping in the DSMP context will be measured by adapting the RCOPE (Pargament, Koenig, and Perez) instrument particularly measuring spiritual coping strategies identified by diabetic individuals. Areas include "I pray to and believe in God", "God keeps me alive", "I turn things over to God", "God changes my unhealthy behaviors", "God supplies my needs", "I read the Bible", and "I ask religious or spiritual individuals help me". The responses will be "1 = Not at all; 2 = Somewhat; 3 = Quite a bit; 4 = A great deal". The higher score reflects better spiritual coping.

CONTACTS AND LOCATIONS:
Overall Officials: Meizi He, PhD, Principal Investigator — The University of Texas at San Antonio
Locations (1):
- Human Nutrition Lab, UTSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available in December 2020.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Sarkar U, Fisher L, Schillinger D. Is self-efficacy associated with diabetes self-management across race/ethnicity and health literacy? Diabetes Care. 2006 Apr;29(4):823-9. doi: 10.2337/diacare.29.04.06.dc05-1615. PMID 16567822
- [Background] van Olphen J, Schulz A, Israel B, Chatters L, Klem L, Parker E, Williams D. Religious involvement, social support, and health among African-American women on the east side of Detroit. J Gen Intern Med. 2003 Jul;18(7):549-57. doi: 10.1046/j.1525-1497.2003.21031.x. PMID 12848838
- [Background] Naderimagham S, Niknami S, Abolhassani F, Hajizadeh E, Montazeri A. Development and psychometric properties of a new social support scale for self-care in middle-aged patients with type II diabetes (S4-MAD). BMC Public Health. 2012 Nov 28;12:1035. doi: 10.1186/1471-2458-12-1035. PMID 23190685
- [Background] Harris J, McGee A, Andrews F, D'Souza J and Sproston K. The national survey of people with diabetes. Prepared for the Healthcare Commission Sept 2007.
- [Background] Lorig K. Outcome measures for health education and other health care interventions. Sage 1996.
- [Background] Yore MM, Bowles HR, Ainsworth BE, Macera CA, Kohl III HW. Single versus multiple item questions on occupational physical activity. Journal of Physical Activity and Health 3(1), 102-111, 2006
- [Background] Norris AE, Ford K, Bova CA. Psychometrics of a Brief Acculturation Scale for Hispanics in a probability sample of urban Hispanic adolescents and young adults. Hispanic Journal of Behavioral Sciences 18:29-38 (abstr), 1996
- See also: Occupational physical activity is evaluated using a single-item question recommended by Behavioral Risk Factor Surveillance System (BRFSS) . — http://www.cdc.gov/brfss/